CLINICAL TRIAL: NCT07350070
Title: TACE Combined With Tislelizumab, Lenvatinib, and Carvedilol for the Treatment of Unresectable Hepatocellular Carcinoma With Cirrhotic Portal Hypertension: A Multicenter, Simon Two-Stage, Single-Arm Study
Brief Title: TACE Combined With Tislelizumab, Lenvatinib, and Carvedilol for Unresectable HCC With Cirrhotic Portal Hypertension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-05
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC; Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — tislelizumab; lenvatinib; Carvedilol

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, single-arm, Simon two-stage design phase II clinical trial, aiming to evaluate the efficacy and safety of the combined TACE with tislelizumab, lenvatinib and carvedilol in the treatment of unresectable hepatocellular carcinoma (uHCC) patients with liver cirrhosis and portal hypertension. The study plans to recruit a total of 78 patients. The optimal two-stage design is adopted: 23 patients will be enrolled in the first stage. If the objective response rate (ORR, based on mRECIST v1.1) does not reach the preset threshold (≤ 11 responses) then the trial will be prematurely terminated; if it reaches (≥ 12 responses), then the second stage will continue with the enrollment of 55 more patients. Finally, if the number of patients achieving response in the total population is ≥ 43, then the scheme is considered effective.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE Combined With Tislelizumab, Lenvatinib, and Carvedilol arm (Experimental): 1. TACE On-demand TACE: Use 1-2 sessions of TACE depending on the tumor condition.
  2. PD-1 inhibitor Tislelizumab 200 mg intravenous infusion, once every 3 weeks
  3. Lenvatinib Formulation: Tablets; Specifications: 4mg/tablet 8mg (for patients weighing less than 60kg) or 12mg (for patients weighing more than 60kg) once daily, taken half an hour after meals (the time of taking the medication should be as consistent as possible), discontinue medication during TACE treatment
  4. Carvedilol Formulation: Tablets; Specifications: 6.25mg/tablet Initial dose is 6.25mg, and the maintenance dose is 6.25mg - 12.5mg/day. For patients with combined arterial hypertension or heart disease, the dose of carvedilol can be further increased to treat non-liver indications.
  Interventions: Drug: TACE Combined With Tislelizumab, Lenvatinib, and Carvedilol

INTERVENTIONS:
Drug: TACE Combined With Tislelizumab, Lenvatinib, and Carvedilol — All the enrolled patients received standard first-line treatment (TACE combined with tiragolumab and lenvatinib) and were additionally treated with carvedilol. The treatment duration of the study was one year. After the end of the treatment, the patients would be evaluated by the researchers to determine whether to continue the treatment or switch to other first-line treatments.

SUMMARY:
In China, the majority of hepatocellular carcinoma (HCC) cases stem from chronic hepatitis B virus (HBV) infection and subsequent cirrhosis, with patients often presenting at the decompensated stage complicated by clinically significant portal hypertension (CSPH). CSPH not only limits treatment options and worsens prognosis but also leads to the frequent exclusion of such patients from pivotal clinical trials, resulting in a lack of high-level evidence for their management. Carvedilol, a non-selective beta-blocker, is a first-line therapy for portal hypertension. Emerging evidence suggests that this drug class may also modulate the tumor microenvironment and enhance the efficacy of immune checkpoint inhibitors.

To address this unmet need, this study aims to explore a novel quadruple-therapy strategy (TACE + tislelizumab + lenvatinib + carvedilol) for the treatment of unresectable HCC with concurrent cirrhotic portal hypertension. The rationale is twofold: while controlling portal hypertension and safeguarding treatment safety, carvedilol may also potentiate immunotherapy by modulating adrenergic signaling, thereby achieving dual benefits of "liver protection" and "anti-cancer" synergy. Utilizing an efficient Simon's two-stage design, this study will conduct a preliminary assessment of the regimen's efficacy and safety with minimal risk, providing essential data to inform future confirmatory research.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most prevalent malignancies worldwide, characterized by high morbidity and mortality rates, and represents a particularly heavy disease burden in China. Notably, unlike in Western countries, the primary etiology of HCC in China is chronic hepatitis B virus (HBV) infection and the resulting cirrhosis. The vast majority of Chinese HCC patients are diagnosed at the decompensated stage of cirrhosis. This condition not only provides the "soil" for tumorigenesis but also leads to a series of life-threatening complications such as portal hypertension, which severely limits treatment options and adversely affects patient prognosis.

HCC patients with underlying HBV-related cirrhosis frequently present with clinically significant portal hypertension (CSPH). Portal hypertension can lead to severe events such as esophageal and gastric variceal bleeding, ascites, and hepatic encephalopathy. Such patients are typically excluded from pivotal clinical trials, resulting in a lack of high-level evidence-based treatment strategies for this subgroup. Currently, there is no global treatment consensus specifically for this special population, creating a significant challenge in clinical decision-making. Regarding the pharmacological management of portal hypertension, non-selective beta-blockers (NSBBs) are the cornerstone therapy. Among them, carvedilol, which blocks both β1- and β2-adrenergic receptors and possesses mild α1-blocking activity, has been proven in multiple randomized controlled trials (RCTs) to effectively reduce the hepatic venous pressure gradient (HVPG) . Both the Chinese Guidelines for the Diagnosis and Management of Cirrhosis and the American Association for the Study of Liver Diseases (AASLD) guidelines, as well as the Baveno VII International Consensus, recommend carvedilol as a first-line agent for the treatment of portal hypertension in cirrhosis.

More intriguingly, recent research suggests that NSBBs may extend beyond their traditional role in lowering portal pressure to directly modulate the tumor microenvironment. Preclinical studies and retrospective analyses indicate that NSBBs (e.g., propranolol) can inhibit multiple pro-oncogenic signaling pathways and alleviate immunosuppression by blocking β2-adrenergic receptors, thereby potentially enhancing the anti-tumor efficacy of immune checkpoint inhibitors (e.g., PD-1/PD-L1 antibodies) and creating a synergistic effect. However, the specific role and clinical value of this effect in HCC remain unknown and urgently require validation through prospective studies.

Based on the above background, this study aims to investigate a novel "quadruple" comprehensive treatment strategy, namely TACE + tislelizumab (a PD-1 inhibitor) + lenvatinib (a targeted agent) + carvedilol (an NSBB), for uHCC patients with concomitant cirrhotic portal hypertension.

The scientific rationale and innovative significance of this design are as follows:

1. It directly focuses on the large yet often trial-neglected population of HCC patients with portal hypertension in clinical practice, exploring an optimal treatment strategy for them.
2. Dual Benefit of "Liver Protection" and "Anti-Cancer": The addition of carvedilol primarily aims to control portal hypertension and prevent severe cirrhosis-related complications (e.g., bleeding), thereby safeguarding patients to safely receive intensive anti-tumor therapy and potentially expanding the patient population eligible for aggressive anti-Cancer": The addition of carvedilol primarily aims to control portal hypertension and prevent severe cirrhosis-related complications (e.g., bleeding), thereby safeguarding patients to safely receive intensive anti-tumor therapy and potentially expanding the patient population eligible for aggressive anti-cancer treatment.
3. Potential "Sensitization" Effect: We hypothesize that carvedilol may enhance the immunotherapeutic efficacy of tislelizumab by modulating adrenergic signaling pathways and improving the tumor immune microenvironment, achieving a synergistic anti-tumor effect where "1+1>2".
4. Exploring a Novel Regimen with Minimal Risk: Given the unknown safety and efficacy profile of this quadruple regimen, this study employs a Simon's two-stage design. This is an efficient and ethical single-arm study design that allows for futility analysis at an early stage. It enables a preliminary assessment of the rationale and potential of this combined strategy with minimal patient exposure risk and resource consumption, providing crucial preliminary evidence for subsequent confirmatory RCTs.

In summary, this study aims to address a pressing clinical challenge and explore an innovative treatment regimen with the multiple potential benefits of "liver protection," "pressure reduction," and "efficacy enhancement." It is anticipated to open new therapeutic avenues for patients with unresectable HCC complicated by cirrhotic portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* At least one radiologically measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (tumor lesion long axis ≥10 mm on CT scan).
* Newly diagnosed hepatocellular carcinoma without any prior treatment for HCC.
* Child-Pugh liver function score ≤ 7.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1.
* Absence of severe organic diseases affecting major organs (e.g., heart, lung, brain).
* Compensated cirrhosis with clinically significant portal hypertension (meeting any one of the following criteria):

  1. Imaging evidence (ultrasound, CT, or MRI) of portosystemic collateral circulation.
  2. Endoscopic evidence of esophageal or gastric varices.
  3. Liver stiffness measurement (LSM) >25 kPa; or LSM 20-25 kPa with platelet count <150×10⁹/L; or LSM 15-20 kPa with platelet count <110×10⁹/L.

Exclusion Criteria:

* Decompensated cirrhosis.
* Concurrent other malignancies or recurrent HCC.
* Any active, known, or suspected autoimmune disease.
* History of allergy to any component of PD-1 inhibitors, lenvatinib, or carvedilol.
* Severe concurrent medical conditions, including asthma, significant cardiac conduction block, and sinus bradycardia.
* Known human immunodeficiency virus (HIV) infection; or active hepatitis (e.g., hepatitis B/C virus infection).
* Presence of tumor thrombus in the inferior vena cava, hepatic vein, or main portal vein.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From the date of enrollment, until the tumor progresses, the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  ORR is defined as the proportion of patients who achieved the best therapeutic response of PR or CR among all the patients enrolled.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From the date of enrollment, until the tumor progresses, the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  PFS is defined as the time from study enrollment to the first occurrence of disease progression.
Overall survival(OS) | From the date of enrollment, until the patient dies, the assessment period can last up to 60 months.
  OS is defined as the time from the start of the study enrollment to death.
Adverse events (AEs) | From the baseline up to 12 months.
  AE is defined as any event that occurs during the treatment period and is not related to the purpose of the treatment which assessed by CTCAE v4.0.
The rate of decompensation of liver cirrhosis | From the date of enrollment, until the patient dies, or the study concludes (whichever occurs first), the assessment period can last up to 60 months.
  The definition of decompensated portal hypertension in liver cirrhosis is the occurrence of clinical events such as upper gastrointestinal bleeding, hepatic encephalopathy, and liver function failure during the treatment period.

OTHER OUTCOMES:
Difference in treatment effect (Hazard Ratio) between participants with emotional disorders versus non-emotional disorders, assessed by the interaction p-value. | From baseline until death, study conclusion, or up to 60 months (whichever occurs first).
  To explore the efficacy difference of the quadruple therapy between pre-defined subgroups. The primary efficacy endpoint (e.g., Progression-Free Survival) will be analyzed separately within each subgroup (emotional disorders vs. non-emotional disorders).

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, Principal Investigator — Tongji Hospital
Locations (7):
- China (7):
  - Clinical Oncology School of Fujian Medical University, Fujian Cancer Hospital, Department of Hepatobiliary and Pancreatic Oncology, Fuzhou, Fujian
  - Department of Hepatobiliary Surgery, The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hubei Province Tahe Hospital, Taihe, Hubei
  - Division of Hepato-Pancreato-Biliary Surgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Organ Transplant Department,Qilu Hospital, Cheeloo College of Medicine, Shandong University,, Jinan, Shandong
  - Shandong First Medical University Affiliated Provincial Hospital, Jinan, Shandong
  - Qingdao University Affiliated Hospital, Qingdao, Shandong